CLINICAL TRIAL: NCT06803121
Title: The Effect of Core Stability Exercises on Idiopathic Scoliosis in Adolescent Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Christine Bahig Shawky Heneen, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004728
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Idiopathic Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional treatment (Active Comparator): It will be consisted of thirty adolescent females with idiopathic scoliosis and will be treated by traditional treatment (traditional exercises and bracing), two sessions per week for three months (24 sessions).
  Interventions: Other: Traditional treatment
- Traditional treatment + Core stability exercises (Experimental): It will be consisted of thirty adolescent females with idiopathic scoliosis and will be treated by traditional treatment (traditional exercises and bracing) in addition to core stability exercises, two sessions per week for three months (24 sessions).
  Interventions: Other: Traditional treatment; Other: Core stability exercises

INTERVENTIONS:
Other: Traditional treatment — Traditional exercises for scoliosis include breathing exercises, posture training, spinal flexibility exercises, stretching exercises for the involved muscles (especially for the concave side of the curve), and general strengthening exercises for the main muscle groups of trunk, pelvis, and shoulder girdle muscles (especially for the convex side of the curve).
Other: Core stability exercises — The CS training program includes local muscle stability training (transverses abdominis, multifidus, and diaphragm), global muscle stability training (oblique abdominal muscles, psoas major, quadratus lumborum, and pelvic floor muscles), global muscle mobility training (rectus abdominis, back extensors, and hamstring muscles), and strength training of the core muscles through the thoracolumbar fascia by maintaining the neutral spine position. Diaphragmatic breathing technique will be used during exercises.
  Arms: Traditional treatment + Core stability exercises

SUMMARY:
To evaluate the efficacy of core stability (CS) exercises on curve magnitude, posture, trunk deformity and quality of life in adolescent females with idiopathic scoliosis.

DETAILED DESCRIPTION:
Scoliosis is a disease in which the spine deviates or rotates laterally from its normal vertical line, and it can cause decreased spinal movement, weakening of muscles near the spine, reduced pulmonary function, respiratory dysfunction, chronic pain, and psychological suffering. Scoliosis can be classified as idiopathic, congenital, neurofibromatosis, and neuromuscular. Among these types of scoliosis, approximately 80% of patients with scoliosis have AIS, which typically occurs around 10 years of age when healthy bone maturation occurs during adolescence. IS is diagnosed when there are no known causes besides spinal deformity involving a lateral curvature with a Cobb angle ≥10°.

Therapeutic approaches for IS include surgical and conservative treatments. Exercise therapy for IS is considered important for maintaining spinal function when the Cobb angle is <20°. Moreover, the effects of core stabilization exercise have been demonstrated recently for alleviating chronic lower back pain in patients, improving performance in athletes, and preventing sports injuries in athletes. Based on this information, core stabilization exercise may be used effectively to improve neuromuscular imbalance, which is the cause of IS. However, studies on the therapeutic effects of using core stabilization exercise in patients with AIS are still lacking.

Accordingly, the objective of this study is to evaluate the efficacy of core stability exercises on curve magnitude, posture, trunk deformity, and quality of life in adolescent females with idiopathic scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* Their ages will be ranged from 10-19 years.
* All adolescent Females will be diagnosed as idiopathic scoliosis with S shape.
* Cobb angle on anterior-posterior radiograph will be used in the assessment of thoracic and lumbar cure of each patient in this study.
* All adolescent females are not under any other treatment method for idiopathic scoliosis.
* Willingness and ability to comply with the study requirements and give informed consent.

Exclusion Criteria:

* Patients with a history of rheumatologic, neuromuscular, cardiovascular, pulmonary, or renal diseases.
* Patients with congenital scoliosis or spinal deformity.
* Patients who had undergone surgical correction of the spine.
* Patients with a tumor.
* Enrollment in any other clinical trial during the time of this trial.

Ages: 10 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Measurement of Cobb angles | 3 months
  Cobb angles on anterior and posterior spine radiographs taken in standing position. The Cobb angle is the angle between two lines, drawn perpendicular to the upper endplate of the uppermost vertebra involved and the lower endplate of the lowest vertebra involved. Once a patient's Cobb angle is determined, the condition can be further classified on its severity scale of mild, moderate, or severe. Cobb angles will be assessed for all adolescent females in both groups A & B before and after treatment.
Measurement of trunk asymmetry in scoliosis | 3 months
  A scoliometer is an instrument that measures trunk asymmetry in scoliosis, or angle of trunk rotation (ATR). It is a small, non-invasive device (essentially a mini-level) that is placed over the spine while a person is in a forward bending position. The scoliometer reading indicates degree of trunk asymmetry (rotation). Generally, an angle of trunk rotation that is less than 5 degrees is insignificant and may not require follow-up. A measurement of 5 to 9 degrees at least warrants reexamination in six months. A measurement of 10 degrees or greater requires radiologic evaluation for Cobb angle measurement.

SECONDARY OUTCOMES:
Trunk appearance perception scale (TAPS) | 3 months
  TAPS includes 3 sets of figures that depict the trunk from 3 viewpoints: looking toward the back, looking toward the head with the patient bending over (Adam's test), and looking toward the front. This last view has two sets of drawings, one for males and one for females. Each drawing is scored from 1 (greatest deformity) to 5 (smallest deformity) and a mean score is obtained by adding the scores for the 3 drawings and dividing by 3.
The Scoliosis research society-22 questionnaire (SRS-22) | 3 months
  The SRS-22 contains 22 questions covering 5 domains: function/activity, 5 items; pain, 5 items; self-perceived body image, 5 items; mental health, 5 items; and satisfaction with treatment, 2 items. The satisfaction scale was not used in the present study. Each item is scored from 1 (worst) to 5 (best). In the present study, the results are expressed as the mean for each domain (total sum of the domain divided by the number of items answered) and the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ahmed Mohamed Awad, PhD, Study Chair — Professor, Cairo university; Afaf Mohamed Mahmoud Botla, PhD, Study Director — Assistant Professor, Cairo university
Locations (1):
- Al Azhar University, Cairo, Egypt